CLINICAL TRIAL: NCT03736395
Title: Scaling up Schoolwide Positive Behavioral Interventions and Supports (SWPBIS) Framework in Rural Settings Through the Idaho Rural Implementation Model
Brief Title: Scaling up Schoolwide Positive Behavioral Interventions and Supports (SWPBIS) in Rural Idaho Schools
Acronym: I-RIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lindsey Turner, Research Professor, Boise State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-CK-BX-0021
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Problem Behavior
Keywords: Behavioral Symptoms; Disruptive Behavior; Schools; School Teachers
MeSH Terms: conditions — Problem Behavior; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: A portion of participating schools will receive the Idaho Rural Implementation Model (I-RIM) intervention, designed to support implementation of schoolwide positive behavioral interventions and supports (SWPBIS). All other participating schools will only receive basic training session about SWPBIS. The process to determine which schools receive the intervention is random. Intervention is at the school level. Outcomes are at the school level, staff level, and student level (anonymous).
Who Masked: Outcomes Assessor
Masking Description: All data collectors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Schools in this condition will be provided a four-day training about Schoolwide Positive Behavioral Interventions and Supports, and bi-yearly feedback about progress monitoring and action planning.
  Interventions: Behavioral: Control
- I-RIM Intervention (Experimental): Schools in this condition will be provided the same basic training as the control condition, plus the elements of the Idaho Rural Implementation Model (I-RIM).
  Interventions: Behavioral: Idaho Rural Implementation Model

INTERVENTIONS:
Behavioral: Idaho Rural Implementation Model — The Idaho Rural Implementation Model (I-RIM) includes several aspects to support implementation of schoolwide positive behavioral interventions and supports (SWPBIS). In the first year, schools will send a staff member to a coaching institute to build internal capacity. Schools will also receive technical assistance (on-site twice per year and virtual support as needed). Schools will also receive statewide professional learning opportunities, through one group meeting per year, and through access to an invitation-only professional learning community.
  Arms: I-RIM Intervention
Behavioral: Control — Schools in this condition will receive a four-day training session about SWPBIS.
  Arms: Control

SUMMARY:
This project will examine the scale-up of Schoolwide Positive Behavior Intervention Supports (SWPBIS), specifically focusing on rural schools in Idaho. The Idaho Rural Implementation Model (I-RIM) is an approach designed to improve SWPBIS implementation in rural schools, via strategies such as capacity-building, regional coordination, online learning modules, and technical assistance. The study uses a cluster randomized design to allocate 40 schools to one of two conditions: control and intervention. Schools in the control condition will receive basic SWPBIS training. Schools in the intervention condition will receive the basic SWPBIS training plus additional I-RIM supports. To assess SWPBIS implementation and outcomes, process and outcome measures will be collected. Outcomes will include school implementation observations, and teacher and staff implementation measures. Student-level outcomes will include behavior, perceived climate, and academic achievement as measured by the standardized state test. Student-level data include those that are part of standard data collection by schools (such as academic outcomes) and will be de-identified by school officials before sending to the researchers for analysis.

DETAILED DESCRIPTION:
The long-term goal of this project is to support rural schools in implementing practices that can improve student safety and social-emotional outcomes, through the use of Schoolwide Positive Behavior Intervention Supports (SWPBIS). Rural schools experience challenges in implementing systems-changes, and the Idaho Rural Implementation Model (I-RIM) is an approach specifically designed to improve SWPBIS implementation in rural schools through strategies such as capacity-building, regional coordination, online learning modules, and technical assistance. These approaches are all designed to meet the unique challenges and strengths of schools in rural settings.

The study uses a cluster randomized design to allocate 40 schools to one of two conditions: control or intervention. Schools in the control condition will receive basic SWPBIS training. Schools in the intervention condition will receive the basic SWPBIS training plus additional I-RIM supports. This trial is designed to address several aims:

Aim 1: To test the impact of the I-RIM intervention on student-level outcomes, including behavioral outcomes, academic test scores, and perceived safety/climate.

Aim 2. To examine whether changes in student outcomes are mediated by school-level improvements in the speed and fidelity with which SWPBIS is implemented.

Aim 3. To identify school-level factors that are associated with SWPBIS implementation (moderators of intervention effectiveness).

At all schools, baseline data collection will begin in early 2019. The intervention will begin in the spring of 2019 with selected elements of the I-RIM intervention (regional meetings, and a coaching institute) for schools in the intervention condition. All schools will begin SWPBIS implementation in the 2019-20 school year, which will continue through the 2020-2021 school year. Data collection points will be identical for schools in both conditions. Primary student outcome measures include data that are already gathered by schools, including: behavioral outcomes including office disciplinary referrals, suspensions, and expulsions; academic test scores; and perceived climate.

ELIGIBILITY:
Inclusion Criteria:

* School is a public school in a rural location in the state of Idaho, serving students in any combination of grades Kindergarten through grade 12.
* Staff work at a school participating in this trial.
* Student attends a school participating in this trial.

Exclusion Criteria:

* None.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in fidelity of school implementation of positive behavioral interventions and supports (PBIS) | Change in school-level implementation score from baseline to 3-year followup
  Change in fidelity of implementation from baseline (spring 2019) to followup (spring 2022) using the Schoolwide Evaluation Tool (SET; Horner et al 2004) to gather observational data about degree of fidelity of implementation on 0-100% scale where 100% is best possible outcome.
Change over time in student disciplinary outcomes | Change from baseline to following school year (Year 2); change from Year 2 to Year 3
  Percentage of students receiving Office Disciplinary Referrals each school year
Change in student academic outcomes | Change from baseline to following school year (Year 2); change from Year 2 to Year 3
  Percentage of students scoring "Advanced" or "Proficient" on state standardized test (Idaho Standards Achievement Test) in English Language Arts and Mathematics
Change in student perceptions of school climate | Change from baseline to 3-year followup.
  Changes in overall scores on school climate surveys. The overall scale score is created by averaging all items, resulting in scores from 1 to 4 with higher overall scores indicating better climate.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Turner, PhD, Principal Investigator — Boise State University
Locations (1):
- Boise State University, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horner RH, Todd AW, Lewis-Palmer T, Irvin LK, Sugai G, Boland JB. The School-Wide Evaluation Tool: A research instrument for assessing school-wide positive behavior support. Journal of Positive Behavior Interventions 6(1):3-12, 2004.
- [Derived] Calvert HG, Fleming CM, Lowe M, Lewis T, Siebert CF, Havlicak A, Anderson N, Castleton T, Turner L. Training and Technical Assistance Increase the Fidelity of Implementation of a Universal Prevention Initiative in Rural Schools: Results from a 3-Year Cluster-Randomized Trial. Prev Sci. 2025 Jan;26(1):56-68. doi: 10.1007/s11121-025-01776-0. Epub 2025 Feb 3. PMID 39899222
- [Derived] Fleming CM, Calvert HG, Turner L. Supporting implementation of universal prevention initiatives in K-12 schools: impacts on fidelity through organizational readiness and team functioning in a cluster-randomized trial. Implement Sci Commun. 2025 Jan 6;6(1):4. doi: 10.1186/s43058-024-00691-9. PMID 39763002
- [Derived] Calvert HG, McQuilkin M, Havlicak A, Lewis T, Turner L. Acceptability, appropriateness, and feasibility of Rural School Support Strategies for behavioral interventions: a mixed methods evaluation over two years of a hybrid type 3 implementation-effectiveness trial. Implement Sci Commun. 2023 Aug 11;4(1):92. doi: 10.1186/s43058-023-00478-4. PMID 37568206